CLINICAL TRIAL: NCT02100501
Title: Prospective Study of Comparison Between the Modified Atkins Diet and Classic Ketogenic Diet for Intractable Childhood Epilepsy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0003
Record Dates: First submitted 2014-03-26; First posted 2014-04-01 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy
Keywords: Seizure control through dietary therapy in pediatric intractable epilepsy patients.
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atkins diet group: pediatric patients diagnosed with intractable epilepsy. Their ages ranged between 1 to 18 years amd indicated to dietary therapy. the targeting number of patients was 53. enrolled patients are assigned to randomly in one of KD group or Atkins group.
- Ketogenic diet group: pediatric patients diagnosed with intractable epilepsy. Their ages ranged between 1 to 18 years amd indicated to dietary therapy. the targeting number of patients was 51. enrolled patients are assigned to randomly in one of KD group or Atkins group.

SUMMARY:
The Ketogenic diet is a now proven, evidence based treatment of refractory epilepsy. the classic ketogenic diet (KD) is based on a ratio of fat to carbohydrate and protein, usually 3:1 or 4:1. Fat is proven long-chain triglycerides. The efficacy of the KD has been proven by many multicenter trials. But, side effects of ketogenic diet therapy is severe. The modified atkins diet (MAD) was designed and investigated at Johns Hopkins Hospital, which aimed to propose a less restrictive dietary treatment that would be more palatable to children and adolescents with less side effects. The MAD consist of a nearly balance diet (60% fat, 30% protein, and 10% carbohydrates by weight), without any restriction on the recommended daily calories. Some literature suggested that the MAD is an effective treatment for refractory epilepsy. But, no randomised controlled study has been tried. the investigators aimed in this prospective study to evaluate the efficacy, safety and tolerability of MAD comparing to KD. The patients were recruited between age 3 to 18 years old with intractable epilepsy. Enrolled patients were randomly assigned to either one of two groups; the KD group and MAD group. The patients were required to attend outpatient clinic after 1, 3month to record their seizure frequency and severity, while their dietary treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 1 to 18 year old patients diagnosed with intractable epilepsy which shows frequency with more than 1 per week, 4 per month even though at least more than 2 antiepileptic drug treatment.

Exclusion Criteria

* Patients heve been tried KD or MAD before.
* Patients with renal stones, hyperlipidemia, cardiologic problems.
* Other conditions not adjust for dietary therapy.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: the patients were recriuted from the Pediatric Neurology Outpatient Clinic, Severance Children's Hospital. This study conducted on 104 (Ketogenic diet - 51, Atkin's diet - 53) patients diagnosed with intractable epilepsy which shows frequency with more than 1 per week, 4 per month even though at least more than 2 antiepileptic drug treatment.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
seizure outcome 3months after dietary therapy. | 3 months
  1 and 3 month after dietary therapy, enrolled patients were required to visit outpatient clinic to record their seizure frequency. we compile statistics and compare seizure frequencies before and after dietary treatment in each KD group and MAD group.

CONTACTS AND LOCATIONS:
Overall Officials: Hoon-Chul Kang, MD, Principal Investigator — Severance Children's Hospital, Yonsei University college of medicine.
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea

REFERENCES:
- [Derived] Kim JA, Yoon JR, Lee EJ, Lee JS, Kim JT, Kim HD, Kang HC. Efficacy of the classic ketogenic and the modified Atkins diets in refractory childhood epilepsy. Epilepsia. 2016 Jan;57(1):51-8. doi: 10.1111/epi.13256. Epub 2015 Dec 10. PMID 26662710